CLINICAL TRIAL: NCT03744767
Title: Adjuvant Anti-Mineralocorticoid-Receptor Treatment in Anti-VEGF Refractory Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr Irmela MANTEL (Other)
Responsible Party: Sponsor-Investigator, Dr Irmela MANTEL, lead consultant, Head of the medical retina service, Principal Investigator, Privatdocent, Eye Hospital Jules Gonin
Organization: Eye Hospital Jules Gonin (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 184/14
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Intervention Model Description: all participants receive fixed monthly intravitreal anti-VEGF injections for 6 months, plus adjuvant treatment during 4 months, followed by 2 months without adjuvant treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single treatment arm (Experimental)
  Interventions: Drug: Spironolactone 50 MG

INTERVENTIONS:
Drug: Spironolactone 50 MG — oral administration of Spironolactone, 25mg daily for 1 week, then 50mg daily until visit Month 3, followed by 25mg daily from visit Month 3 to visit Month 4

SUMMARY:
Prospective, non-comparative, mono-center pilot study. Patients with neovascular age-related macular degeneration (nAMD), responding insufficiently to the maximal standard care with monthly intravitreal anti-VEGF injections are given adjuvant oral mineralocorticoid receptor antagonists for 4 months and observed for any changes in vision or retinal structure during the 4 months of adjuvant treatment, plus 2 additional months without adjuvant treatment.

DETAILED DESCRIPTION:
Hypothesis Systemic anti-Mineralocorticoid-Receptor treatment may be a valuable adjuvant treatment in anti-VEGF refractory nAMD, potentially allowing for better absorption of the exudative fluid.

Aim To estimate the effect of systemic anti-Mineralocorticoid-Receptor treatment on eyes with nAMD which have remained exudative despite monthly anti-VEGF treatment for at least 6 months prior to enrolment.

Objectives Primary objective

* To calculate the changes induced in retinal thickness following adjunct systemic anti-Mineralocorticoid-Receptor treatment Secondary objective
* To calculate the changes induced following adjunct systemic anti-Mineralocorticoid-Receptor treatment in the following ocular parameters

  * Thickness of the neuro-retina (foveal)
  * Amount of subretinal fluid (foveal and highest elevation)
  * Height of retinal pigment epithelium detachment (foveal and highest elevation)
  * Central (Subfoveal) choroidal thickness, and at 500um nasal and temporal to the fovea
  * Presence / absence of exudative signs on OCT, according to the type of fluid (intraretinal cysts, subretinal fluid)
  * Best corrected visual acuity (number of letters)

Medications:

Standard medical treatment (monthly intravitreal injections with anti-VEGF) will be continued during this trial, no current medications will be altered. The medication spironolactone, an MR antagonist will be added to the currently prescribed medications (phase IV). The standard dose of 50mg once daily per os will be prescribed for 3 months (first week 25mg only for treatment introduction and safety), tapered during month 4 (25mg once daily).

In the case of a patient current taking a medication with contra-indications for this drug, then the conflicting medication will be exchanged for an equivalent treatment option, where this is not possible then these patients will be excluded from the study. The patient will be withdrawn from the study in case of any serious side effects attributable to spironolactone (increased K+ above 5.5mmol/l).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neovascular age-related macular degeneration, as confirmed on angiography by a retinal specialist (IM or AA)
* Aged more than 50 years (inherent to AMD)
* Unresponsive to maximal (monthly) anti-VEFG treatment (Ranibizumab or Aflibercept) for at least 6 months: persistant intra- or subretinal fluid on spectral domain optical coherence tomography at each visit 1 month after last injection.
* Treatment with anti-VEGF for nAMD for at least 12 months
* No contra-indications for adjunctive Spironolactone treatment

Exclusion Criteria:

* Confounding retinal pathology eg. myopic chorioretinopathy, diabetic retinopathy, vascular occlusion, retinal dystrophy and other retinal pathology
* Polypoidal choroidal vasculopathy
* Vitreomacular traction
* Poor quality OCT (image quality does not allow the grading / measures on OCT)
* High arterial pressure (>160/100)
* K+>5.0 mmol/l at baseline
* Na+ <135 mmol/l at baseline
* Creatinine clearance under 30mL/min (calculation : coefficient*(140-age)*weight/creatinine in the serum; coefficient = 1.23 for males and 1.04 for females)
* Acute renal failure
* Renal dialysis
* Non-specified renal problem
* Arrhythmia
* Cardiovascular comorbidity with thromboembolic risk
* Known hypersensitivity to Spironolactone
* Ongoing medication with eplerenone (Inspra®)
* Decompensated hepatic cirrhosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2015-09-22 (Actual); Study Completion 2015-09-22 (Actual)

PRIMARY OUTCOMES:
Retinal thickness change | Month 3, Month 6
  retinal thickness in micrometers measured from the internal limiting membrane (ILM) to Bruch's membrane on optical coherence tomography

SECONDARY OUTCOMES:
Best-corrected visual acuity | Month 3, Month 6
  on ETDRS chart
central retinal thickness | Month 3, Month 6
  automatic values from SD-OCT after segmentation correction, in micrometers
central retinal volume | Month 3, Month 6
  automatic values from SD-OCT after segmentation correction
foveal retinal thickness | Month 3, Month 6
  manual measurement in micrometers from ILM to Bruch membrane at the fovea
maximum neuroretinal thickness with cystic changes | Month 3, Month 6
  manual measure in micrometers from ILM to outer segments of photoreceptors
subretinal fluid thickness | Month 3, Month 6
  manual measure in micrometers between outer segment layer and pigment epithelium
pigment epithelium detachment height | Month 3, Month 6
  manual measure in micrometers from the RPE layer to Bruch's membrane
subfoveal choroidal thickness | Month 3, Month 6
  manual measure in micrometers on enhanced depth OCT imaging

IPD SHARING:
Plan to Share IPD: Undecided